CLINICAL TRIAL: NCT04969172
Title: A Phase II Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Exosomes Overexpressing CD24 to Prevent Clinical Deterioration in Patients With Moderate or Severe COVID-19 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eli Sprecher, MD (Other Government)
Collaborators: OBCTCD24 Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Eli Sprecher, MD, Dr. Guy Choshen, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0206-21-TLV
Record Dates: First submitted 2021-07-18; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Disease
Keywords: AE- Adverse event; BUN - Blood urea nitrogen; CI- Confidence Interval; CMP - Clinical monitoring plan; CONSORT- Consolidated Standards of Reporting Trials; CRF - Case Report Form; DAMP- Damage-associated molecular patterns; DMEM- Dulbecco's Modified Eagle's Medium; GCP - Good Clinical Practice; GMP- Good Manufacturing Practice; GVHD- Graft-versus-host disease; HCT - Hematopoietic stem cell transplantation; ICH- International Conference on Harmonization; IDSA- Infectious Diseases Society of America; IRB- Institutional Review Board; ITT- Intend-to-Treat analysis set; mITT- Modified Intent-to-Treat analysis set; NLR - Neutrophil-to-lymphocyte ratio; PCR - Polymerase chain reaction; PI- Principal Investigator; PP- Per-Protocol analysis set; SA- Safety analysis set; SAE- Serious adverse event; SoA- Schedule of Activities; TLR- Toll-like receptors
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: A Phase II Randomized, double-blind, Placebo-controlled Study to Evaluate the safety and efficacy of exosomes overexpressing CD24 to prevent clinical deterioration .The study population will include patients with moderate or severe COVID-19 infection and laboratory markers predictive of the cytokine storm from the Corona department of each site, who have provided an informed consent.
Who Masked: Participant, Investigator
Masking Description: 155 patients will be randomized in a 2:1 ratio to receive either 1010 exosome particles -103 patients, or placebo- 52 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1010 Exosome (Active Comparator): 103 patients will receive either 1010 exosome particles.
  Interventions: Drug: Exosomes overexpressing CD24
- Placebo (Placebo Comparator): 52 patients will receive placebo- saline.
  Interventions: Drug: Exosomes overexpressing CD24

INTERVENTIONS:
Drug: Exosomes overexpressing CD24 — The suggested therapeutic agent here is based on an existing therapeutic platform that uses exosomes that were engineered to overexpress CD24 that can directly suppress the cytokine storm. The exosomes will be isolated and purified from human embryonic kidney T-REx™-293 cells that constitutively express high levels of human CD24.

SUMMARY:
A Phase II Randomized, double-blind, Placebo-controlled Study to Evaluate the safety and efficacy of exosomes overexpressing CD24 to prevent clinical deterioration .The study population will include patients with moderate or severe COVID-19 infection and laboratory markers predictive of the cytokine storm from the Corona department of each site, who have provided an informed consent.

155 patients will be randomized in a 2:1 ratio to receive either 1010 exosome particles (103 patients) or placebo (52 patients).The exosomes will be diluted in 4ml normal saline for inhalation, administered once daily (QD) for 5 days.

Placebo (saline) will be prepared for inhalation and administered in the same manner as the exosomes.

DETAILED DESCRIPTION:
The exosomes will be diluted in 4ml normal saline for inhalation, administered once daily (QD) for 5 days.

Placebo (saline) will be prepared for inhalation and administered in the same manner as the exosomes.

Study treatments will be given as add-on to standard of care. Following the 5 days of treatment, patients will remain in follow-up for 23 additional days. Patients who will be discharged before the end of the 5-day treatment period will continue to receive treatment at home. Treatment administration and the study assessments will be carried out by the research personnel at the home of the patient, implementing the required protective measures.

On Day 28, when the isolation period is completed, these patients will arrive at the study site for the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. A COVID-19 diagnosis confirmed with a SARS-coV-2 viral infection positive polymerase chain reaction (PCR) test
2. Age 18-80 years
3. Severity of disease according to the following criteria (at least one clinical parameter and one laboratory parameter are required):

   a. Clinical and Imaging-based evaluation i. Respiratory rate > 23/min and < 30/min ii. SpO2 at room air ≤94% and ≥90% iii. Bilateral pulmonary infiltrates >50% within 24-48 hours or a severe deterioration compared to imaging at admission b. Evidence of an exacerbated inflammatory process i. LDH score> 450 U/L ii. CRP >50 mg/L iii. Ferritin >1650 ng/ml iv. Lymphocytes >800 cells/mm3 v. D-dimers >1 mcg/ml
4. Willing and able to sign an informed consent

Exclusion Criteria:

1. Age<18 years or >80 years
2. Any concomitant illness that, based on the judgment of the Investigator is terminal
3. Ventilated patient
4. Pregnancy (positive urine pregnancy test [women of childbearing potential only]) or breastfeeding
5. Patients with Immunodeficiency (eg, CLL, HIV, rituximab therapy)
6. Unwilling or unable to provide informed consent
7. Participation in any other Interventional study in the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2021-07-11 (Actual); Primary Completion 2022-07-11 (Estimated); Study Completion 2022-07-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of EXO-CD24 in the treatment of patients with moderate or severe COVID-19 disease | One year
To assess the efficacy of EXO-CD24 in the clinical improvement of COVID-19 disease | One year
To evaluate respiratory failure (defined as the need for mechanical ventilation, ECMO, non-invasive ventilation, or high-flow oxygen devices) rate. | One year
To evaluate the death rate. | One year
To evaluate time to improvement and recovery (COVID-19 clinical severity score of 3 or lower). | One year
To evaluate time from hospitalization to hospital discharge. | One year
To assess the COVID-19-related symptoms using patient-reported outcome measure (PRO) score. | One year

SECONDARY OUTCOMES:
To evaluate the effect of EXO-CD24 on the respiratory rate. | One year
To evaluate the effect of EXO-CD24 on the change in blood oxygen saturation (SpO2). | One year
To evaluate the effect of EXO-CD24 on the proportion of patients requiring ventilation. | One year
To evaluate the effect of EXO-CD24 on the level of inflammatory markers (eg, CRP, ferritin, fibrinogen, di-dimers, IL-6, LDH, lymphocytes count. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pala M, Yilmaz SG. Circular RNAs, miRNAs, and Exosomes: Their Roles and Importance in Amyloid-Beta and Tau Pathologies in Alzheimer's Disease. Neural Plast. 2025 Apr 8;2025:9581369. doi: 10.1155/np/9581369. eCollection 2025. PMID 40235521